CLINICAL TRIAL: NCT02431676
Title: Trial of Behavioral Weight Loss and Metformin Treatment to Lower Insulin Growth Factor in Cancer Survivors
Brief Title: Survivorship Promotion In Reducing IGF-1 Trial
Acronym: SPIRIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Maryland Cigarette Restitution Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: J14148; IRB00035653 (Other: JHMIRB)
Record Dates: First submitted 2015-04-21; First posted 2015-05-01 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Prostate Cancer; Lung Cancer; Colon Cancer; Melanoma of Skin; Endometrial Cancer; Liver Cancer; Pancreatic Cancer; Rectal Cancer; Kidney Cancer; Other Solid Malignant Tumors
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Colonic Neoplasms; Melanoma; Endometrial Neoplasms; Liver Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Kidney Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Self-Directed (Active Comparator): In this group, the study staff will meet with you once at the beginning of the study to give you written information about weight management.
  Interventions: Behavioral: Self-control weight loss
- Coach Directed Behavioral Weight Loss (Experimental): The Remote Lifestyle Coaching intervention is based on the Call Center Directed intervention to help you loss weight
  Interventions: Behavioral: Coach Directed Behavioral Weight Loss
- Metformin (Experimental): This group will be given the study drug called Metformin. Metformin comes in tablet form that you take with meals
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Participants will receive metformin, an oral medication for type 2 diabetes.Participants randomized to the metformin intervention will receive metformin up to 2,000 mg per day.Dosing can be flexible, two or three times per day with meals as tolerated for 12 months.
  Arms: Metformin
Behavioral: Coach Directed Behavioral Weight Loss — Behavioral-based telephonic coaching with web-based support to promote healthy lifestyle and weight loss in overweight and obese adults.The goal of this intervention is to achieve at least 5% weight loss in the first six months of the intervention and maintain these improvements through month twelve by meeting dietary and exercise goals
  Arms: Coach Directed Behavioral Weight Loss
Behavioral: Self-control weight loss
  Arms: Self-Directed

SUMMARY:
This is a prospective, single-center randomized trial with three arms, and an allocation ratio of 1:1:1. The study design is an efficacy study to evaluate the effect of metformin and coach-directed behavioral weight loss versus self-directed weight loss on insulin-like growth factor (IGF)-1 and IGF-1 to THE IGFBP-III ratio blood levels after 6 and 12 months of intervention. The coach-directed Behavioral Weight Loss arm is a web-based remote delivery and communication system that promotes healthy behavioral changes. The Metformin arm is a pharmaceutical intervention of oral metformin. This is a secondary prevention study for men and women who have survived solid malignant tumors

ELIGIBILITY:
Inclusion Criteria:

* Women and men ages 18 or older
* Have been previously diagnosed with a malignant solid tumor, completed their required surgical, and/or chemotherapy and/or radiation curative intent therapy at least three months prior to enrollment, and have an anticipated treatment-free life span of 12 months or longer. Chemoprophylaxis with tamoxifen or aromatase inhibitors for breast cancer in women and anti- Luteinizing hormone-releasing hormone (LHRH) therapy for prostate cancer in men will be permitted.
* Have a BMI of 25 kg/m^2 or greater and weight <=400 lbs.
* Willingness to accept randomization to each of the three arms
* Willingness to change diet, physical activity, and weight
* Regular access to computer with a reliable Internet connection
* Ability to send and receive emails
* Ability to complete online forms
* Access to phone
* Willingness to provide written informed consent

Exclusion Criteria:

* Women who are breastfeeding, pregnant, or planning pregnancy within the next year
* Medication-treated diabetes
* Fasting blood glucose >=200 mg/dL, or fasting blood glucose >=126 and <200 mg/dL and HbA1C >=7%
* Current or prior regular use of metformin within the past 3 months
* Uncontrolled concurrent medical condition likely to limit compliance with the study interventions
* Received any chemotherapy (unless anti-hormonal therapy) and/or radiation three months or less prior to the proposed intervention date
* Have a prior history of lactic acidosis by self-report
* Prior or planned bariatric surgery
* Have significant renal disease or dysfunction defined as Estimated glomerular filtration rate (eGFR)<45
* Have significant hepatic dysfunction [Aspartate aminotransferase (AST)/Alanine transaminase (ALT) ≥ 2 x upper limit of normal (ULN) or reported liver disease]
* Self-reported average consumption of > 14 alcoholic drink per week
* Currently enrolled or planned to enroll in weight loss program
* Hemoglobin <9 g/dl
* Platelet count <100
* White blood cell count (WBC) <2.5
* Plans to relocate from the area within one years
* Use of prescription weight loss medication(s) (e.g., lorcaserin, topiramate/phentermine, phentermine, liraglutide, and bupropion/naltrexone), including off label use of drugs for weight loss or over-the-counter weigh loss medications such as Orlistat within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Yeh, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins ProHealth, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tilves C, Yeh HC, Maruthur N, Juraschek SP, Miller E, White K, Appel LJ, Mueller NT. Increases in Circulating and Fecal Butyrate are Associated With Reduced Blood Pressure and Hypertension: Results From the SPIRIT Trial. J Am Heart Assoc. 2022 Jul 5;11(13):e024763. doi: 10.1161/JAHA.121.024763. Epub 2022 Jun 22. PMID 35730613
- [Derived] Tilves C, Yeh HC, Maruthur N, Juraschek SP, Miller ER, Appel LJ, Mueller NT. A behavioral weight-loss intervention, but not metformin, decreases a marker of gut barrier permeability: results from the SPIRIT randomized trial. Int J Obes (Lond). 2022 Mar;46(3):655-660. doi: 10.1038/s41366-021-01039-2. Epub 2022 Jan 6. PMID 34987204
- [Derived] Hu JR, Yeh HC, Mueller NT, Appel LJ, Miller ER 3rd, Maruthur NM, Jerome GJ, Chang AR, Gelber AC, Juraschek SP. Effects of a Behavioral Weight Loss Intervention and Metformin Treatment on Serum Urate: Results from a Randomized Clinical Trial. Nutrients. 2021 Jul 31;13(8):2673. doi: 10.3390/nu13082673. PMID 34444833
- [Derived] Mueller NT, Differding MK, Zhang M, Maruthur NM, Juraschek SP, Miller ER 3rd, Appel LJ, Yeh HC. Metformin Affects Gut Microbiome Composition and Function and Circulating Short-Chain Fatty Acids: A Randomized Trial. Diabetes Care. 2021 Jul;44(7):1462-1471. doi: 10.2337/dc20-2257. Epub 2021 May 18. PMID 34006565
- [Derived] Juraschek SP, Plante TB, Charleston J, Miller ER, Yeh HC, Appel LJ, Jerome GJ, Gayles D, Durkin N, White K, Dalcin A, Hermosilla M. Use of online recruitment strategies in a randomized trial of cancer survivors. Clin Trials. 2018 Apr;15(2):130-138. doi: 10.1177/1740774517745829. Epub 2018 Jan 24. PMID 29361843

RESULTS

PARTICIPANT FLOW:
Groups:
- Self-Directed: In this group, the study staff will meet with you once at the beginning of the study to give you written information about weight management.
  Self-control weight loss
Period: Overall Study
Arm/Group | Self-Directed | Coach Directed Behavioral Weight Loss | Metformin
Started | 40 | 39 | 42
Completed | 40 | 38 | 40
Not Completed | 0 | 1 | 2
Not completed — no lab obtained | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Directed | Coach Directed Behavioral Weight Loss | Metformin | Total
Number analyzed (Participants) | 40 | 39 | 42 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (8.5) | 60.9 (9.7) | 59.5 (9.0) | 59.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 32 | 96
  Male | 8 | 7 | 10 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 18 | 17 | 20 | 55
  Other non-black races | 22 | 22 | 22 | 66
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.7 (4.9) | 35.5 (5.0) | 35.0 (6.3) | 35.0 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: IGF-1 Levels
Description: Insulin-like growth factor (IGF)-1 levels (ng/ml) at 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Self-Directed | Coach Directed Behavioral Weight Loss | Metformin
Number analyzed (Participants) | 40 | 38 | 40
ng/ml | 73.2 (19.9) | 73.6 (20.9) | 71.2 (21.4)

2. Secondary Outcome: IGF-1 Levels
Description: IGF-1 at 12 months
Time Frame: 12 months
Population: Data was obtained for 39 participants in the self-directed arm, 37 in the coach directed arm and 37 in the metformin arm for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Self-Directed | Coach Directed Behavioral Weight Loss | Metformin
Number analyzed (Participants) | 39 | 37 | 37
ng/ml | 73.4 (20.7) | 76.6 (25.7) | 76.2 (25.7)

3. Secondary Outcome: IGF-1 to IGFBP3 Level Ratio (Molar Ratio)
Description: IGF-1 level to IGFBP3 level ratio (molar ratio) at 6 months.
Time Frame: 6 months
Population: Data was obtained for 39 participants in the self-directed arm, 37 in the coach directed arm and 36 in the metformin arm for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Self-Directed | Coach Directed Behavioral Weight Loss | Metformin
Number analyzed (Participants) | 39 | 37 | 36
ratio | 0.18 (0.047) | 0.18 (0.065) | 0.17 (0.046)

4. Other Pre Specified Outcome: Weight Measured by Scale(Kg)
Description: Changes in weight among Metformin group, or coach-directed Groups versus the self-directed arm at 6 and 12 months
Time Frame: 6 and 12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Body Mass Index Measured by Scale and Tap(kg/m2)
Description: Changes in BMI among Metformin arm, or coach-directed behavioral weight loss arm versus the self-directed arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: EuroQol Score Assessed by Questionnaire
Description: Changes in EuroQol score among Metformin arm, or coach-directed behavioral weight loss arm versus the self-directed arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Dietary Intake Assessed by Questionnaire
Description: Changes in dietary intake among Metformin arm, or coach-directed behavioral weight loss arm versus the self-directed arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Physical Activity Amount Assessed by Questionnaire
Description: Changes in physical activity amount among Metformin arm, or coach-directed behavioral weight loss arm versus the self-directed arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Fasting Glucose Levels
Description: Changes in fasting glucose among Metformin arm, or coach-directed behavioral weight loss arm versus the self-directed arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Insulin Levels
Description: Changes in insulin among Metformin arm, or coach-directed behavioral weight loss arm versus the self-directed arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Hemoglobin A1C Levels
Description: Changes in Hb-A1C among Metformin arm, or Coach-directed behavioral weight loss arm versus the Self-control weight loss arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Interleukin (IL)-6 Levels
Description: Changes in IL-6 among Metformin arm, or coach-directed behavioral weight loss arm versus the self-directed arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Interleukin 8 Levels
Description: Changes in IL-8 among Metformin arm, or coach-directed behavioral weight loss arm versus the self-directed arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: C-reactive Protein (CRP) Levels
Description: Changes in CRP among Metformin arm, or coach-directed behavioral weight loss arm versus the self-directed arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Side Effects Assessed by Side Effect Questionnaire
Description: assessing side effect among Metformin arm, or coach-directed behavioral weight loss arm versus the self-directed arm at 6 and 12 months.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 month
Arm/Group | Self-Directed | Coach Directed Behavioral Weight Loss | Metformin
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39 | 0/42
Serious Adverse Events (participants affected / at risk) | 5/40 | 5/39 | 12/42
Other Adverse Events (participants affected / at risk) | 10/40 | 3/39 | 6/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Self-Directed (N=40) | Coach Directed Behavioral Weight Loss (N=39) | Metformin (N=42)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
CVD (Cardiac disorders) | 0 | 0 | 3
Other (General disorders) | 3 | 3 | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Self-Directed (N=40) | Coach Directed Behavioral Weight Loss (N=39) | Metformin (N=42)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Heart Disease (Cardiac disorders) | 0 | 0 | 2
Injury (Musculoskeletal and connective tissue disorders) | 5 | 1 | 2
Gallstone (Gastrointestinal disorders) | 2 | 0 | 0
Gallstone removal (Surgical and medical procedures) | 2 | 0 | 0
bariatric surgery (Surgical and medical procedures) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT02431676/Prot_SAP_000.pdf